CLINICAL TRIAL: NCT02241174
Title: Efficacy of 0.005% Sodium Hypochlorite Final Rinse Solution on the Reduction of Staphylococcus Aureus Colonization in Atopic Dermatitis: A Randomized Controlled Trial
Brief Title: 0.005% Sodium Hypochlorite Final Rinse Solution in Atopic Dermatitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study materials have expired, no patients were enrolled
Sponsor: Makati Medical Center (Other)
Responsible Party: Principal Investigator, Jamaine Cruz, MD, Dr., Makati Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SodiumHypochloriteAD
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Hypochlorite (Experimental): The 0.005% sodium hypochlorite solutions will be prepared from the commercially available Clorox® at 6% solution. 0.83ml of the 6% sodium hypochlorite solution will be taken and incorporated to a-100ml absolute distilled water.
  Interventions: Drug: Sodium Hypochlorite
- Placebo (Placebo Comparator): 100ml distilled water will be used as a placebo and will be stored on amber bottles identical with the treatment group
  Interventions: Drug: Sodium Hypochlorite

INTERVENTIONS:
Drug: Sodium Hypochlorite — The 0.005% sodium hypochlorite solutions will be prepared from the commercially available Clorox® at 6% solution. 0.83ml of the 6% sodium hypochlorite solution will be taken and incorporated to a-100ml absolute distilled water. This 100ml solution will be stored in an amber glass bottle at room temperature unexposed to light at a maximum of 23 months

SUMMARY:
This study will determine the safety and efficacy of diluted bleach bath solution as final rinse on the reduction of Staphylococcus aureus colonization among children and adult Filipinos with mild to moderate atopic dermatitis..

DETAILED DESCRIPTION:
Objective: To determine the safety and efficacy of 0.005% sodium hypochlorite final rinse solution on the reduction of Staphylococcus aureus colonization among children and adult Filipinos with mild to moderate atopic dermatitis.

Design: Randomized, double blind, controlled clinical trial. Setting: Makati Medical Center, Dermatology Outpatient Department Participants: Patients with mild to moderate atopic dermatitis, seen at Makati Medical Center Dermatology Outpatient Department.

Sample size: 68 (34 treatment group, 34 placebo group) Intervention: Eligible patients will be randomly allocated to two groups. The subjects will either be in the treatment group (0.005% sodium hypochlorite) or in the placebo group (bath water). Subjects will use a liter of 0.005% sodium hypochlorite as a final rinse solution during bathing for the treatment group and a liter of bath water for the placebo group. This intervention will be done twice a week for 12 weeks. Both patients and assessors will be blinded to the treatment assignments.

Assessment of Outcome: The outcomes will be assessed at weeks 4 and 12. Primary outcome measure will use culture findings, physician's global assessment (PGA) of severity of disease and eczema area and severity index (EASI) score. Secondary outcome measure will assess adverse effects during follow-up at weeks 4 and 12.

Data Analysis: Kruskal-Wallis Test will be used to compare the significant difference in scores between the two groups and Wilcoxon Signed Rank Test will be used to compare significant difference of before and after scores within each group.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females more than 8 years old.
2. Subjects with clinical diagnosis of atopic dermatitis (based on Hannifin and Rajka criteria).
3. Healthy subjects with no other skin disease.
4. Subjects without any prior topical or oral antibiotic two weeks prior to the enrollment period. Those who had undergone course of topical and oral antibiotic are given at least 2 weeks washout period.

Exclusion Criteria:

1. Severe Atopic dermatitis requiring hospitalization.
2. Hospitalized and debilitated patients.
3. Subjects with other serious skin disorder, pigmentation or extensive scarring in affected areas.
4. Subjects who have a known history or clinically relevant allergy, in particular to chlorine containing compounds.
5. Pregnant women and nursing mothers.
6. Subjects who are in a situation, which, in the opinion of the investigator, may interfere with optimal participation in the study.
7. Subjects participating or having participated in a clinical trial within 1 month before enrollment in the study.
8. Subjects who cannot communicate with the investigator (>18 years old) or are unaccompanied by parent or legal guardian (<18 years old).
9. Subjects who are unable to follow-up.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Culture and sensitivity findings | 12 weeks
  The primary outcome of interest is the reduction of S. aureus colonization in skin lesion and the clinical improvement at week 4 and week 12.
Eczema Assessment Severity Index (EASI) | 12 weeks
  Clinical decrease in the disease severity of atopic dermatitis Eczema Assessment Severity Index (EASI) b. Clinical decrease in the disease severity of atopic dermatitis Eczema Assessment Severity Index (EASI)
  Body regions to be assessed:
  1. Head/Neck
  2. Upper extremities
  3. Trunk
  4. Lower extremities
  In each of the body areas, the following key signs will be assessed:
  1. Erythema (E)
  2. Induration (I)
  3. Excoriation (Ex)
  4. Lichenification (L)
  Scoring from the above features:
  1. 0 - none
  2. 1 - mild
  3. 2 - moderate
  4. 3 - severe
  Body Surface Area involvement score:
  1. 0 = no eruption
  2. 1 = <10%
  3. 2 = 10%-29%
  4. 3 = 30% - 49%
  5. 4 = 50% - 69%
  6. 5 = 70% - 89%
  7. 6 = 90% - 100%
  EASI Score Body region EASI Score Head/neck (E + I + Ex + L) x Area x 0.1 Upper extremities (E + I + Ex + L) x Area x 0.2 Trunk (E + I + Ex + L) x Area x 0.3 Lower extremities (E + I + Ex + L) x Area x 0.4 EASI Sum of above scores
Physician Global Assessment (PGA) Scale | 12 weeks
  Severity of disease at baseline
  Mild:
  Moderate:
  Severe:
  Rating scale for PGA of Clinical Response at the end of the treatment
  Rating % Improvement Week 4 Week 12
  Cleared 100%
  Excellent improvement 90-99%
  Marked improvement 75-89%
  Moderate improvement 50-74%
  Slight improvement 30-49% No appreciable improvement 0-29%

SECONDARY OUTCOMES:
Adverse Effect | 12 weeks
  An adverse effect is an adverse event for which the causal relation between the intervention and the event is at least a reasonable possibility. The term 'adverse effect' applies to all interventions, while 'adverse drug reaction' (ADR) is used only with drugs. Both will be measured in the study. All subjects will be asked if they have experienced any untoward effects from the intervention. In the event that any adverse events and adverse effects will be noted, immediate medical attention will be given to the participant(s) and the expenses of which, will be shouldered by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Marie L. Sarrosa, MD, FPDS, Principal Investigator — Makati Medical Center; Jamaine Melisse L Cruz, MD, Principal Investigator — Makati Medical Center
Locations (1):
- Makati Medical Center, Makati, NCR, Philippines